CLINICAL TRIAL: NCT00776360
Title: The Effect of Oxytocin on Gastric Emptying in Patients With Gastro Paresis
Brief Title: The Effect of Oxytocin on the Gastric Emptying
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Bodil Ohlsson, Department of Clinical Sciences, Division of Internal Medicine, Skane University Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 29/2008
Record Dates: First submitted 2008-10-17; First posted 2008-10-21 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Postprocedural Delayed Gastric Emptying
Keywords: oxytocin; gastroparesis; diabetics; The effect of oxytocin on gastric emptying
MeSH Terms: conditions — Gastroparesis | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oxytocin, gastric emptying (Experimental): Oxytocin is given to study the gastric emptying rate
  Interventions: Drug: oxytocin
- oxytocin (Placebo Comparator): sodium chloride is given to study gastric emptying rate
  Interventions: Drug: oxytocin

INTERVENTIONS:
Drug: oxytocin — 80mIE/min as continuous infusion for 70 minutes
  Other Names: syntocinon
Drug: oxytocin — 80 mU/ min of oxytocin infusion for 70 min along with measuring the gastric emptying by ventricle scintigraphy
  Other Names: syntocinon

SUMMARY:
The investigators are going to examine whether oxytocin has a prokinetic effect on gastric emptying in patients suffering from gastro paresis. Oxytocin infusion will be compared with sodium chloride infusion.

DETAILED DESCRIPTION:
The investigators are going to examine whether oxytocin has a prokinetic effect on gastric emptying in patients suffering from gastro paresis. Oxytocin infusion will be compared with sodium chloride infusion.The gastric emptying is estimade by sitntigraphy during 70 minutes, and performed twicw. Once with saline and once with oxytocin.

ELIGIBILITY:
Inclusion Criteria:

* Gastroparesis in diabetics

Exclusion Criteria:

* Treatment with other prokinetics, other severe organic or psychological diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To examine whether oxytocin improves gastric emptying in gastroparesis | dec 2008-dec 22009